CLINICAL TRIAL: NCT03287583
Title: Pilot Randomized Control Trial of an SBIRT Intervention for Gambling
Brief Title: SBIRT Intervention for Gambling Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Christopher Welsh, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00067608
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: participants will be randomized to receive either the Gambling Specific SBIRT Intervention or enhanced control.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT (Experimental): SBIRT intervention for Gambling
  Interventions: Behavioral: SBIRT for Gambing
- Control (Other): Participants randomized to the enhanced control condition will receive a handout with gambling resources.
  Interventions: Other: Enhanced Control

INTERVENTIONS:
Behavioral: SBIRT for Gambing — The SBIRT intervention uses a brief gambling screening assessment to determine whether or not a participant is at risk for problem gambling. This is followed by a structured short brief intervention to assist people in better understanding their risk for gambling and what they can do to limit that risk.
  Arms: SBIRT
Other: Enhanced Control — Participants randomized to the enhanced control condition will receive a handout with gambling resources.
  Arms: Control

SUMMARY:
Disordered gambling, like substance misuse, has been associated with various medical problems and adverse health outcomes. The Maryland Center of Excellence on Problem Gambling, along with experts in the fields of disordered gambling and behavior change, will work with the Maryland State Department of Health and Mental Hygiene's Behavioral Health Administration to develop a problem gambling-specific Screening, Brief Intervention and Referral to Treatment (SBIRT) intervention targeting individuals receiving medical care in general primary care clinics. The investigators will evaluate the feasibility and acceptability of inserting the problem gambling intervention in to preexisting substance use SBIRT services being provided in clinics in the state. In addition, the investigators will establish a clinic prevalence for gambling and finally, conduct a randomized trial using the problem gambling SBIRT intervention to see if it is effective in helping patients reduce their problematic gambling behaviors.

DETAILED DESCRIPTION:
The Substance Abuse and Mental Health Services Administration (SAMHSA) has made health care and health systems integration one of its main priorities to ensure that behavioral health is consistently incorporated within the context of health care delivery systems. However, this initiative has been focused on substance use disorders and mental health disorders that have not included gambling disorder. Disordered gambling (DG) is highly associated with substance use disorders, severe mental illness, depression, domestic violence and suicide. Disordered gambling has also been linked with adverse health conditions and behaviors. Morasco et al., in their analysis of data from the National Epidemiologic Survey of Alcohol and Related Conditions (NESARC), found that persons with DG were more likely to have a range of medical problems including tachycardia, angina, cirrhosis or other liver disease. Even moderate levels of gambling along with more severe levels of DG have been associated with adverse health consequences and unhealthy life style factors. Morasco et al. report that at risk gamblers (defined as gambling five or more times in the past 12 months) who they estimate compose 25% of the population, were more likely to have experienced a severe injury in the past year, receive emergency room treatment, have hypertension, be obese, have histories of mood, anxiety, alcohol use and nicotine use disorders. In a more recent study, Black et al. found individuals with DG were at higher risk for chronic medical conditions including obesity, heartburn/stomach conditions, headaches, head injury with loss of consciousness, sleep disorders, mood/emotional concerns, and anxiety, tension or stress. Individuals in the DG group also were more likely to have poorer health habits. They were more likely to avoid exercise, to drink alcohol while pregnant, smoke greater than or equal to a pack of cigarettes per day to drink or more servings of caffeine a day and to watch or more hours of television weekly. Subjects meeting DG criteria in this study were also less likely to have regular dental check-ups and more likely to delay medical care for financial reasons. Additionally the DG subjects were more likely to have at least one emergency room visit and at least one hospitalization for mental health reasons in the past year.

Individuals with gambling problems have been found to utilize medical and behavioral health services at higher rates.

Studies have also reported significant rates of gambling and problem gambling in primary care settings. Pasternak and Fleming in a study of patients in primary care, that 80% had gambled and 6.2% met criteria for problem gambling (score of 3 or more on South Oaks Gambling Screen, SOGS). Additionally they report that gambling disorder was even more prevalent among nonwhites and those from lower socioeconomic groups. In a study of individuals receiving free or reduced-cost dental care, Morasco & Petry found rates of problem gambling to be significantly higher than the general population. In their sample, among those receiving disability, 26% met criteria for disordered gambling and among those not receiving disability 14% met criteria based on SOGS scores. Other studies have found prevalence rates of gambling problems of between 3 and 5% in primary care settings. However, these studies did not include any frequency of gambling items nor an explanation of the range of behaviors meant by "gambling" and have not included the less severe "at risk" gamblers. This study will also address the need to improve the effectiveness of DG screening strategies in actual clinical practice and to effectively identify not just those individuals who are exhibiting multiple symptoms of gambling disorder but those fall into an "at risk" level of gambling that has been associated with multiple poor health outcomes.

A prevalence study conducted in Maryland supports the likelihood of significant health issues among those who are identified as at risk, problem or disordered gamblers. This study found that 90% of adults in Maryland had gambled in their lifetimes. Over 21% had gambled at least monthly in the past 12 months which would fit the definition of at risk gambling group that compromised 25% of the subjects in the NESARC study who presented increased medical issues and utilization. Those who had ever gambled as well the at risk and problem gambling groups in the Maryland survey also reported higher levels of health risk behaviors (i.e. higher alcohol intake, more frequent drug use, daily smoking) and reported poorer health status. The rates of problem/pathological gambling for all adults was found to be 3.4% and at risk gambling 9%. African Americans(17.3%) were found to have a significantly higher rate of at risk as well as problem and disordered gambling compared to other ethic/racial groups (10.2% white, 11.7% other ethnic/racial combined). The lowest socioeconomic group was also found to have the highest rates of problem/pathological gambling (15%). Therefore, conducting gambling specific screening and brief intervention in these high risk groups within Maryland is strongly indicated.

While the research as sited above clearly indicates that individuals who are experiencing gambling related harms in their lives are likely to experience higher rates of medical and behavioral health problems and utilize health care services, they are not necessarily likely to seek specific help for gambling problems. Strikingly, Kessler et al. reported that while nearly half of their large national sample who met criteria for lifetime gambling disorder received treatment for mental health or substance use disorders, none had received any specific treatment for gambling problems. Indeed, it is estimated that only between 1 to 3% of individuals nationwide who meet criteria for gambling disorder access gambling specific treatment services.While this is in part due to internal factors in individuals with gambling disorder such as desire to resolve problems on their own, shame, guilt and denial, there are also provider/institutional factors that are significant. Primary among these is the absence of screening for gambling problems.

Screening, Brief Intervention and Referral to Treatment (SBIRT) is an evidence based, public health approach for delivery of early intervention services in medical and primary care settings for individuals at risk for or experiencing substance use disorders. The most extensive research evidence for the effectiveness of this approach has been with those presenting indicators of alcohol abuse. Additionally Brief interventions (BI) have been found to be effective for a range of non-alcohol substance abuse issues. While many studies have demonstrated that brief interventions with disordered gamblers are effective, these studies have not focused on identifying or providing brief interventions in actual clinical or primary care settings. Research has suggested that there are considerable clinician as well as client factors that contribute to reluctance to address the topic of gambling practice. To our knowledge no study has sought to obtain both client and clinician input into the content and process feasibility of providing screening and intervention for risk for GD in real clinical settings to address clinician and client concerns.

Both research and treatment provider surveys have demonstrated that only a very small percentage of individuals who experience gambling related harms are likely to seek treatment. Furthermore, there is evidence that at risk gamblers who may comprise 20-25% of the adult population are likely to experience increase levels of health related problems and utilize health care services at higher rates than non/low-risk gamblers. However, has been little to no research on how to effectively screen for risk for gambling in health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Attending the recruitment clinic at University of Maryland
* English Speaking

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
gambling time back follow-up | one month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, SMART clinic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided